CLINICAL TRIAL: NCT01573039
Title: Definition of Cut Off for PCR - Quantitative and Antigenemia in the Diagnosis of Cytomegalovirus (CMV) Disease in Serum-positive Kidney Transplant Recipients
Brief Title: Cut Off for the Diagnosis of Cytomegalovirus (CMV) Disease in Serum-positive Kidney Transplant Recipients
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CAPPesq 0045/11
Record Dates: First submitted 2012-04-04; First posted 2012-04-06 (Estimated); Last update posted 2014-04-04 (Estimated); Status verified 2013-01

CONDITIONS: Cytomegalovirus Disease
Keywords: Kidney transplantation; PCR quantitative; cytomegalovirus; antigenemia
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
CMV disease is a challenge to the success of renal transplantation. Recently, the investigators analyzed data from 792 renal transplant recipients performed at our hospital between 1999 and 2005. After the usual exclusions, 663 patients were analyzed. This population showed that the incidence of CMV disease is stable and occurs in approximately 20-22% of all patients and invasive disease in approximately 5% every year. In seronegative patients and those receiving anti-lymphocyte (AL), CMV prophylaxis, done with ganciclovir for 90 days is our routine and in the majority of transplant centers. In seropositive patients without associated risk factors (such as the use of AL) universal prophylaxis is not done. Rather, in this group, early diagnosis, by detection of antigenemia or viremia by quantitative PCR, is performed in patients who show symptoms compatible with CMV disease. In the investigators analysis the incidence of CMV disease in seropositive patients is around 16%. These patients are usually hospitalized and treated with GCV IV for 14-21 days. This leads to an additional costs of admissions, biopsies for the diagnosis of disease invasion, etc. Besides these costs, the survival of the grafts in the long run is lower in patients with CMV disease than in those without CMV, particularly when associated with acute rejection. In recent years, monitoring of viremia (PCR / antigenemia) and preemptive treatment when it reaches substantial values, have increasingly been suggested. Patients in whom the detection of viremia in progressive values is detected would be treated as outpatients before the disease develops. To turn this hypothesis into reality, there is an urgent need to define cutoff values for CMV-PCR in the detection of developing CMV disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 14 years and younger than 75 years
* Seropositive for CMV (IgG)
* Kidney transplant recipients

Exclusion Criteria:

* Patients who received anti-lymphocyte induction
* Patients with organ transplants double

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Kidney transplant recipients
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2011-11; Primary Completion 2012-11 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Establish a cutoff for viremia, antigenemia detected by PCR and quantitative-to event for CMV disease. | Day 0,7,14,21,28,35,42,56,63, 70,77,84,91,98, 105,112,120

CONTACTS AND LOCATIONS:
Overall Officials: Elias David-Neto, MD, Principal Investigator — University of Sao Paulo General Hospital
Locations (1):
- Hospital das Clinicas - Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo, Brazil